CLINICAL TRIAL: NCT03917576
Title: Heart Rate Changes in Response to an Exercise Test and to a High Intensity Interval Training Session in Subjects With Normoglycaemic, Prediabetes, and Type 2 Diabetes Mellitus State
Brief Title: Heart Rate During Exercise in Type 2 Diabetes
Acronym: HRinT2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Los Lagos (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RP010317
Record Dates: First submitted 2019-04-07; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes Mellitus; Hyperglycemia; Heart Rate; Exercise Training
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: We will compare a type 2 diabetes mellitus group during exercise, with another hyperglicaemic, and normoglicaemic group in the heart rate maxymum.
Who Masked: Investigator
Masking Description: The exercise session consisted of 1-minute cycling at high intensity (workload during each interval was set at ~80-100 % maximal power (i.e., load in Watts) achieved during the incremental exercise test with a workload that allowed to work until the volitional muscle failure in 1-minute), followed by 2-minutes of inactive resting period (sitting still on the cycle ergometer), and was repeated 10 times (1x2x10 protocol; 1:2:10 to work:rest:repetitions respectively). The exercise session was supervised individually by exercise professionals, monitoring the heart rate with a continuous telemetric heart rate sensor (Polar FT4, PolarTM, Finland). During the single HIIT session, the HR pre each interval (HR-preINT) and the HR post each interval (HR-postINT) of cycling was recorded individually. In addition, we calculated and report the percentage of maximum heart rate in each interval, delta of HR increment and delta HR recovery for each 10-interval HIIT are reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoglicamic group (Active Comparator): Control normoglycaemic participants
  Interventions: Other: Exercise training intervention
- Hyperglicaemic group (Active Comparator): Control hyperglicaemic group
  Interventions: Other: Exercise training intervention
- Experimental group (Experimental): Experimental Type 2 Diabetes Mellitus Group
  Interventions: Other: Behavioral

INTERVENTIONS:
Other: Behavioral — The resting heart rate (HRrest), maximum HR (HRmax), HR recovery (HRRTEST), delta HR recovery (ΔHRRTEST) were measured by continuous telemetric heart rate sensor (Polar FT4, PolarTM, Finland) during an incremental exercise test designed to obtain maximum oxygen consumption (VO2max) on a cycle ergometer (Lode Corival, Groningen, The Netherlands) similar with previous studies using similar cohort. An indirect calorimetry/ergospirometry system (Ultima CPXTM metabolic system, Medgraphics, Minnesota, USA) was used to measure VO2max until volitional exhaustion. Thus, the modified Astrand volitional protocol was applied in the participants of all NG, Pre-T2D and T2D groups increasing the load (i.e., Watts) 25 W each 2 min to women, and 50 W each 2 min to men.
  Other Names: Incremental exercise test
  Arms: Experimental group
Other: Exercise training intervention — Subjects also participated in a single HIIT session composed of 10-cycling intervals, using a Lode Corival cycle ergometer. The exercise session consisted of 1-minute cycling at high intensity (workload during each interval was set at ~80-100 % maximal power achieved during the incremental exercise test with a workload that allowed to work until the volitional muscle failure in 1-minute), followed by 2-minutes of inactive resting period (sitting still on the cycle ergometer), and was repeated 10 times (1x2x10 protocol; 1:2:10 to work:rest:repetitions respectively).
  Other Names: Exercise training intervention with HIIT
  Arms: Hyperglicaemic group; Normoglicamic group

SUMMARY:
Exercise training is a cornerstone for the prevention and treatment of metabolic disorders and associated cardiometabolic complications such as type 2 diabetes mellitus (T2D) and hypertension. Similar to the beneficial health effects after performing conventional continuous exercise modalities, high intensity interval training (HIIT) has been reported as an effective alternative exercise-modality to improve glucose homeostasis in both prediabetes subjects and individuals with T2D diagnosed. In this regard, although multiple HIIT-based interventions commonly report acute and long term benefits on body composition, cardiorespiratory fitness and insulin sensitivity in metabolically compromised subjects, little is known about the acute cardiovascular response (i.e., at heart rate level) during HIIT in subjects with different glucose control.

HIIT is described as performing brief periods of exercise at vigorous or maximal intensity, interspersed with inactive or low intensity recovery phases of variable duration. In order to characterize different HIIT-based protocols, exercise intensity is usually defined as relative percentages of individual maximal cardiorespiratory fitness (VO2max) or relative maximal power output values. Nevertheless, the need for specific technological equipment to assess these parameters usually limit the prescription and recommendations of HIIT in clinical settings and other public health contexts at massive level. Additionally, the use of self-perceived exertion scales and heart rate (HR) variations upon HIIT have been demonstrating to be accessible and feasible strategies to regulate exercise intensity during HIIT. For example, it was reported that HR and self-perceived exertion scores increased progressively in T2D subjects, parallel to the oxygen consumption rate throughout an acute HIIT session performed on cycle ergometer. Consequently, it is conceivable to hypothesize that determining HR variations during HIIT might optimize the recommendation of this training methodology in metabolically compromised subjects as those at risk or with T2D diagnosed. Therefore, the aim of the present study was To describe and compare the acute heart rate changes in response to an incremental maximal exercise test and a single HIIT session between normoglycaemic (NG), prediabetes (Pre-T2D) and type 2 diabetes mellitus (T2D) subjects.

DETAILED DESCRIPTION:
This cross-sectional study will use a non-probabilistic sample of 75 adult subjects, characterized as healthy normoglycaemic and others with disturbed glucose homeostasis subjects, all referred by a physician to the exercise programme of our research centre. The present study will be carried out in accordance with the Declaration of Helsinki and was approved by the Scientific Ethics Committee of the Universidad de La Frontera. All volunteers read and signed an informed consent. The inclusion criteria will be; a) aged 18-60 y; b) previously screened by physician professional; c) diagnosed with normoglycaemic, prediabetes or T2D state; d) and living in Temuco city. The exclusion criteria will be; a) low maximal cardiorespiratory fitness (defined as VO2max ≤21 ml/kg-1/min-1) below the expected value for the subject's sex and age 11; b) not receiving pharmacologic hypotensive treatment with β-blockers; and c) having no musculoskeletal limitations to perform exercise cycling. The total sample size will be divided in three groups according to the standard glycaemic classification 12; normoglycaemic (NG, n = 32), pre-diabetes (Pre-T2D, n = 30) and type 2 diabetes (T2D, n = 13). The study considered three stages of measurements (enrollment, exercise test, single HIIT session).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 y
* previously screened by physician professional
* diagnosed with normoglycaemic, prediabetes or T2D state
* living in Temuco city

Exclusion Criteria:

* low maximal cardiorespiratory fitness (defined as VO2max ≤21 ml/kg-1/min-1) below the expected value for the subject's sex and age
* not receiving pharmacologic hypotensive treatment with β-blockers
* having no musculoskeletal limitations to perform exercise cycling

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
Maximum heart rate | 12 weeks
  Measured before and after 12 weeks of high-intensity interval training

SECONDARY OUTCOMES:
Resting heart rate | 12 weeks
  Measured before and after 12 weeks of high-intensity interval training
Heart rate pre each HIIT-interval | 12 weeks
  Measured before and after 12 weeks of high-intensity interval training
Heart rate post each HIIT-interval | 12 weeks
  Measured before and after 12 weeks of high-intensity interval training

CONTACTS AND LOCATIONS:
Locations (1):
- Cristian ALvarez, Osorno, Chile

IPD SHARING:
Plan to Share IPD: No
We hope to send data of individual participant according with requirements by e-mail.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03917576/Prot_SAP_000.pdf